CLINICAL TRIAL: NCT00374335
Title: Multiple Hemangiomas and Large Cutaneous Hemangiomas of Infancy: Incidence of Hepatic Hemangiomatosis
Brief Title: Incidence of Hepatic Hemangiomatosis in Patients With Cutaneous Hemangiomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: Medical College of Wisconsin (Other); University of California, San Francisco (Other); Columbia University (Other); Baylor College of Medicine (Other); Northwestern University (Other); St. Justine's Hospital (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 06 02 029E
Record Dates: First submitted 2006-09-07; First posted 2006-09-11 (Estimated); Results first posted 2011-09-12 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Hemangioma
Keywords: prospective cohort study
MeSH Terms: conditions — Hemangioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- infants with cutaneous hemangiomas (Other)
  Interventions: Procedure: abdominal ultrasound; Other: Dermatologic Examination

INTERVENTIONS:
Procedure: abdominal ultrasound — abdominal ultrasound to detect hepatic hemangiomas
Other: Dermatologic Examination — Complete dermatologic examination

SUMMARY:
This study will attempt to determine how common liver hemangiomas are in children with infantile hemangiomas by comparing liver ultrasound results in patients with 1-4 cutaneous hemangiomas, 5 or more cutaneous hemangiomas, or at least 1 large hemangioma versus ultrasound results in children without hemangiomas. Other objectives of the study include identifying specific risk factors in patients who have liver hemangiomas and identifying risk factors in children with symptomatic liver hemangiomas.

DETAILED DESCRIPTION:
Hemangioma of infancy is the most common tumor of childhood occurring in 4% to 10% of infants. While most hemangiomas are benign in behavior and involute spontaneously, some can cause significant morbidity due to their location and size. In addition, some hemangiomas may be associated with extracutaneous hemangiomas that result in significant morbidity. Certain "high risk" hemangiomas of infancy, specifically multiple cutaneous hemangiomas or a solitary large hemangioma, have been associated with hepatic hemangiomatosis; however, the exact number or size of the cutaneous lesions at which the risk increases and the protocol for evaluating these patients remain controversial. The true prevalence of hepatic hemangiomatosis is unknown since there have been no large scale prospective studies evaluating clinically asymptomatic patients with cutaneous hemangiomas for the presence of hepatic hemangiomatosis.

One of the primary objectives of this study is to determine the incidence of hepatic hemangiomatosis in patients with hemangiomas of infancy by comparing hepatic ultrasound imaging results of patients with 1-4 cutaneous hemangiomas, 5 or more cutaneous hemangiomas, or at least 1 large hemangioma >30 cm2 versus imaging results in patients without cutaneous hemangiomas. The study will also attempt to identify specific risk factors associated with the development of hepatic hemangiomatosis and to identify associated risk factors in patients with clinically symptomatic hepatic hemangiomatosis.

ELIGIBILITY:
Inclusion Criteria:

* Infants less than 6 months of age
* clinical diagnosis of 1-4 cutaneous hemangiomas
* clinical diagnosis of 5 or more cutaneous hemangiomas
* clinical diagnosis of at least 1 large cutaneous hemangioma greater than 30 cm2

Exclusion Criteria:

* Infants greater than 6 months of age

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 261 (Actual)
Dates: Start 2006-09; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Drolet, MD, Principal Investigator — Medical College of Wisconsin; Maria Garzon, MD, Principal Investigator — Columbia University; Kimberly A Horii, MD, Principal Investigator — Children's Mercy Hospital Kansas City; Denise Metry, MD, Principal Investigator — Baylor College of Medicine; Sarah Chamlin, MD, Principal Investigator — Northwestern University-Children's Memorial Hospital; Ilona J Frieden, MD, Principal Investigator — University of California, San Francisco; Julie Powell, MD, Principal Investigator — St. Justine's Hospital; Anne Lucky, MD, Principal Investigator — Children's Hospital of Cincinnati; Eulalia Baselga, MD, Principal Investigator — Hospital de la Santa Crue i Santa Pau
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Chiller KG, Passaro D, Frieden IJ. Hemangiomas of infancy: clinical characteristics, morphologic subtypes, and their relationship to race, ethnicity, and sex. Arch Dermatol. 2002 Dec;138(12):1567-76. doi: 10.1001/archderm.138.12.1567. PMID 12472344
- [Background] Boon LM, Burrows PE, Paltiel HJ, Lund DP, Ezekowitz RA, Folkman J, Mulliken JB. Hepatic vascular anomalies in infancy: a twenty-seven-year experience. J Pediatr. 1996 Sep;129(3):346-54. doi: 10.1016/s0022-3476(96)70065-3. PMID 8804322
- [Background] Metry DW, Hawrot A, Altman C, Frieden IJ. Association of solitary, segmental hemangiomas of the skin with visceral hemangiomatosis. Arch Dermatol. 2004 May;140(5):591-6. doi: 10.1001/archderm.140.5.591. PMID 15148105
- [Background] Hughes JA, Hill V, Patel K, Syed S, Harper J, De Bruyn R. Cutaneous haemangioma: prevalence and sonographic characteristics of associated hepatic haemangioma. Clin Radiol. 2004 Mar;59(3):273-80. doi: 10.1016/S0009-9260(03)00267-8. PMID 15037141
- [Background] Bruckner AL, Frieden IJ. Hemangiomas of infancy. J Am Acad Dermatol. 2003 Apr;48(4):477-93; quiz 494-6. doi: 10.1067/mjd.2003.200. PMID 12664009
- [Derived] Horii KA, Drolet BA, Baselga E, Frieden IJ, Metry DW, Morel KD, Newell BD, Nopper AJ, Garzon MC; Hemangioma Investigator Group. Risk of hepatic hemangiomas in infants with large hemangiomas. Arch Dermatol. 2010 Feb;146(2):201-3. doi: 10.1001/archdermatol.2009.391. No abstract available. PMID 20157038

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Cutaneous Hemangiomas (multiple > 5, 1-4, or at least 1 hemangioms >30 cm2)
Period: Overall Study
Arm/Group | Group 1
Started | 261
Completed | 261
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 261
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 261
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.3 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192
  Male | 69
Region of Enrollment [Number; unit: participants]
  United States | 232
  Spain | 13
  Canada | 16

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Hepatic Hemangiomas Identified on Abdominal Ultrasound
Description: The number of participants with cutaneous infantile hemangiomas (1-4 cutaneous hemangiomas, greater than 5 cutaneous hemangiomas, or at least one large cutaneous hemangioma) who were found to have hepatic hemangiomas on abdominal ultrasound
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 261
participants | 24

2. Secondary Outcome: Risk Factors Associated With the Development of Hepatic Hemangiomas
Description: Which participants with cutaneous infantile hemangiomas (1-4 cutaneous hemangiomas, greater than 5 cutaneous hemangiomas, or at least 1 large cutaneous hemangioma) were found to have hepatic hemangiomas on abdominal ultrasound
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 261
participants | 24

3. Primary Outcome: Presence of Hepatic Hemangiomas on Abdominal Ultrasound
Description: as for outcome 1
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/261
Other Adverse Events (participants affected / at risk) | 0/261

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No